CLINICAL TRIAL: NCT04556916
Title: Early Detection of Prostate Cancer by Liquid Biopsy
Brief Title: Early Detection of Prostate Cancer
Acronym: PROLIPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0014; 2019-A02253-54 (Other: IDRCB)
Record Dates: First submitted 2020-06-23; First posted 2020-09-21 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; liquid biopsy; circulating tumour cells
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men over 40 being suspicious of prostate cancer (Experimental): Per patient 49 ml of peripheral blood sample after signing consent and performing before the 1st prostate biopsy
  Interventions: Diagnostic Test: Blood sample
- Men over 40 with no suspicion of prostate cancer (Experimental): Per patient 49 ml of peripheral blood sample after signing consent
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Per patient 49 ml of peripheral blood sample :
  * 21ml divided into 3 TransFix or EDTA 7ml tubes will be sent to Hamburg for subsequent CTCapture analysis;
  * 28ml divided into 4 EDTA 7ml tubes will be sent to Montpellier for subsequent EPIDROP analysis (21 ml), PHI analysis (7 ml) and plasma isolation.

SUMMARY:
This study is the early detection of prostate cancer by analysing circulating bloodbased biomarkers. Based on our latest developments, we primarily aim to assess the validity of CTCs (circulating tumour cells) and tumour cell products circulating in blood (DNA, exosomes) for early PCa (Prostate cancer) detection.

In the first discovery period, the investigators will assess which Liquid biopsy marker will provide the best discrimination between the patients with histologically proven PCa and age-matched noncancer controls. Further subset analysis with special emphasis on the identification of high risk PCa patients with aggressive tumours as defined by a Gleason score ("gold standard") of 8 or higher (ISUP 4 and higher), will be performed. The resulting biomarker candidates will then be further explored in the subsequent training and validation study (years 2 and 3) in order to obtain the single blood test or combination of tests with the highest sensitivity and specificity for detection of early PCa and/or high-risk PCa. The investigators will also compare these new biomarkers with recently FDA cleared CE-IVD assays for early detection of prostate cancer, based on classic peripheral tumour markers, such as Prostate Health Index (PHI) and PCA3. Follow up evaluations will be initiated to assess the prognostic relevance of the candidate biomarkers determined in this project. Here, the investigators will set up the data management system including all relevant information on the tissues collected and the results of the analyses as well as the clinical data of the patients investigated in this study.

DETAILED DESCRIPTION:
In this preclinical validation study patients suspicious of prostate cancer who will undergo initial prostate biopsy are going to be asked for blood samples during a routine visit. Each patient will have had an MRI (Magnetic Resonance Imaging) as part of the care before performing the biopsy. The investigators will draw a total of 49 ml peripheral blood from consented patients before the initial diagnostic biopsy is taken. Within this project, validation of liquid biopsy assays for early detection of prostate cancer patients is the primary goal.

In order to determine CTC numbers, 21 ml of blood will be subjected to either CTC-Capture, and 28 ml for the EPIDROP analysis according to standard protocol (For analysis of circulating blood products plasma, analysis of tumor specific mutations or promotor methylation, analysis of extracellular vesicles and microRNA). The investigators will also analyze the Prostate Health Index marker from the additional EDTA tube (7 ml).

The investigators will assess whether CTC counts and/or detection of tumor specific blood products will provide discrimination between the men with histologically proven prostate cancer and agematched non-cancer controls as well as identification of high-risk PCa patients.

Furthermore, the investigators will compare results from tested liquid biopsy assay with current standard of early prostate cancer detection using both serum PSA and digital rectal examination, MRImp and PSA density.

The discovery phase is a non-blind study on 70 subjects with elevated PSA, and 50 negative controls (Healthy patients no suspicion of prostate cancer; PSA<2.5). The 70 patients are patients with suspected prostate cancer and will undergo prostate biopsy.

The samples will be tested for the 3 biomarkers (CTCs, cfDNA, exosome). The validation study is a non-blind study on 167 subjects with elevated PSA and designated for a biopsy (this biopsy may be positive (presence of cancer) or negative (no cancer revealed by the biopsy)), and 33 negative controls. The samples will be tested with the best biomarkers or biomarker combination selected in the discovery phase.

ELIGIBILITY:
Inclusion Criteria Patient :

* Men over 40 being suspicious of prostate cancer
* Subject with PSA ≥ 4 and designated for biopsy
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures
* mpMRI done before prostate biopsy
* Subject must be covered by public health insurance
* Signed informed consent form

Inclusion Criteria Subject Control Patient patient free from prostatic disease :

* Men over 40 with no suspicion of prostate cancer
* Subject with PSA < 2.5 and normal digital rectal examination
* Subject must be covered by public health insurance
* Signed informed consent form

Exclusion Criteria Patient :

* Subject with histologically confirmed prostate cancer
* Subject with a verified viral infection (HIV or Hepatitis)
* Subject under Finasteride treatment
* Subject under hormonal treatment (analogs, antagonists, androgenics)
* Subject with other cancer diagnosed
* Subject unable to sign consent
* Planned longer stay outside the region that prevents compliance with the visit plan
* Subject deprived of liberty, protected adults or vulnerable persons
* Urinary infection ≤ 2 months
* Subject excluding health insurance registration
* Subject refusing to perform prostate biopsy
* Subject who are in a dependency or employment with the sponsor or the investigator

Exclusion Criteria Subject Control :

* Subject with histologically confirmed prostate cancer
* Subject with a verified viral infection (HIV or Hepatitis)
* Subject under Finasteride treatment
* Subject with other cancer diagnosed
* Subject unable to sign consent
* Planned longer stay outside the region that prevents compliance with the visit plan
* Subject deprived of liberty, protected adults or vulnerable persons
* Urinary infection ≤ 2 months
* Subject excluding health insurance registration

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men over 40 years
Enrollment: 320 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2033-09-15 (Estimated)

PRIMARY OUTCOMES:
Discovery of CTCs and tumour cell products circulating in blood (DNA, exosomes) for early PCa detection. | Expected duration of the recruitment of the discovery phase: 12 months
  Evaluate Liquid biopsy marker between the patients with histologically proven PCa and age-matched noncancer controls.

SECONDARY OUTCOMES:
Detection duration of the recruitment of the validation study. | Expected duration of the recruitment of the validation study: 24 months
  The most marker(s) assay(s) will be further explored in the subsequent training and validation study in order to obtain the blood test to detect early prostate cancer in patients with elevated serum PSA.
Validity of blood test with the highest specificity for detection of early PCa and/or high-risk PCa. | Expected duration of the recruitment of the validation study: 24 months
  Combination of complementary circulating biomarkers as liquid biopsy of cancer (CTCs, circulating tumor DNA & exosomes).
Validity of blood test with the highest specificity for detection of early PCa and/or high-risk PCa. | Expected duration of the recruitment of the validation study: 24 months
  Measure the prognostic relevance of candidate biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Catherine ALIX-PANABIERES, MCU-PH, Principal Investigator — University Hospital, Montpellier
Locations (4):
- France (4):
  - CHU Montpellier - Département d'urologie et transplantation rénale, Montpellier
  - CHU Montpellier - Laboratoire des Cellules Circulantes Rares Humaines, Montpellier
  - Clinique Beau Soleil - Service d'urologie, Montpellier
  - CHU de Nîmes - Service Urologie Andrologie Sexologie, Nîmes

IPD SHARING:
Plan to Share IPD: No